CLINICAL TRIAL: NCT03595033
Title: iPad Application Based Therapy Intervention in School Age Children With Surgically Treated Hydrocephalus
Brief Title: Hydrocephalus iPad-App Based Intervention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIN_HCPiPad_001
Record Dates: First submitted 2018-05-29; First posted 2018-07-23 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Hydrocephalus; Hydrocephaly; Hydrocephalus in Children
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Phase (Experimental): Throughout the intervention phase, participants will attend weekly intervention visits. During these visits, an occupational therapist (OT) will educate the participant and their caregiver on the therapy plan which includes the iPad apps to be completed during the week. The participants will be asked to complete their therapy plan for 1 hour per day at home, 4 days per week.
  Interventions: Device: iPad app-based intervention

INTERVENTIONS:
Device: iPad app-based intervention — The 1-hour of home based intervention will break into three 20-min sessions, each including iPad apps targeting one of the three domains of deficits: visual attention, visual-spatial reasoning, and visual-motor skills.

SUMMARY:
This is a pilot study examining the feasibility and efficacy of using Apple iPad applications ("apps") during therapy interventions that target visual motor, visual attention, and visual-spatial reasoning skills in school age children who were previously treated surgically for hydrocephalus. Each subject will participate in an initial assessment and baseline MRI, followed by 6-weeks of iPad app-based interventions, and finally a follow-up assessment and a follow-up MRI.

DETAILED DESCRIPTION:
Long term visuospatial and visuomotor functional deficits are common in pediatric patients with surgically treated hydrocephalus. The deficits are often mild/moderate at early school age although the gap may widen as the children grow older, leading to increasing adverse impact on school performance and academic achievement. The proposed study will generate initial pilot data for the usage of iPad application based therapy intervention for the treatment of cognitive deficits common to pediatric hydrocephalus. It will help determine the optimal intensity and duration of training protocol adapted for the study. In addition, the sensitivity of neuroimaging (DTI) in response to the therapy will be assessed and validated as a biomarker that reflects the neuroanatomical alterations underpinning the outcome changes. This study will generate the crucial data to support the design of future Phase III clinical trial with the long term goal as changing the current standard of care in order to prevent neurocognitive and sensorimotor deficits before the injury to neural circuitry becomes irreversible.

The participants who meet the inclusion criteria and do not opt-out of participation will be called by a study coordinator to ensure eligibility and to schedule the initial assessment date. Participation in this study will include 8-10 study visits. These visits include 2 neuropsychological assessments, 2 MRI visits, and 6 weekly visits during intervention phase. MRI visit can be combined with the neuropsychological assessment visit if possible at both the pre- and post intervention time points.

ELIGIBILITY:
Inclusion Criteria:

* Children, aged 6 to 17 years, with hydrocephalus who have had a surgical intervention
* Deficits in 2 of more of the following neuropsychological testing categories: visual motor, visual attention, or visual reasoning.

Exclusion Criteria:

* Shunt revision within the past one year
* MRI-sensitive programmable shunt or any other MRI-sensitive implant
* Braces or other dental hardware that would interfere with the quality of MRI images (participants with braces are only excluded from the MRI portion of the study)
* Intellectual disability: IQ < 70
* Deficits in one or none of the three following neuropsychological testing categories: visual motor, visual attention, or visual reasoning
* Age 18 years or greater
* Non-English speaking: We will not enroll non-English speaking participants because the iPad applications are not readily available in other languages. All neuropsychological testing materials are also in English.

Ages: 6 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2015-11-24 (Actual); Primary Completion 2018-12-28 (Actual); Study Completion 2018-12-28 (Actual)

PRIMARY OUTCOMES:
General intellectual functioning, including visual-spatial reasoning | Initial assessment and Follow-up assessment (6-8 weeks after Initial assessment)
  The Perceptual Reasoning Index (PRI) of the revision of the Wechsler Abbreviated Scale of Intelligence (WASI-II). PRI includes the subtests Block Design and Matrix Reasoning. The Raw scores of the subtests are converted to T-scores, which are summed for a Sum of T-scores for Perceptual Reasoning. The Sum of T-scores for Perceptual Reasoning is converted to a Composite Score of the PRI, which can be used to find the Percentile Rank. The Block Design raw scores range from 0-51 and the Matrix Reasoning raw scores range from 0-23. The T-score ranges are from 20-54. The Composite Scores range from 40-160.The higher the scores of the subtests, the higher the score on the PRI, the greater the subject's ability to analyze and synthesize abstract visual stimuli and the subject's fluid intelligence, broad visual intelligence, classification and spatial ability, knowledge of part-whole relationships, simultaneous processing, and perceptual organization.
Basic visual perception, visual-motor integration, and graphomotor skills | Initial assessment and Follow-up assessment (6-8 weeks after Initial assessment)
  The Beery-Buktenica Developmental Test of Visual Motor Integration 6th Edition (Beery VMI). The composite score is the sum of the scores of three subtests: Visual-Motor Integration, Visual Perception, and Motor Coordination. The scores for the subtests are calculated using pre-formatted tables to determine the standard score, scaled score, and percentile based off of the raw score. The composite score has a mean of 100 and a standard deviation of 15 for all ages groups, and are based on the means of raw score distribution. The higher the score, the higher the percentile, the greater the subject's ability for visual perception, visual motor-integration, and graphomotor skills.
Visual-spatial processing | Initial assessment and Follow-up assessment (6-8 weeks after Initial assessment)
  The Arrows subtest of the revision of A Developmental Neuropsychological Assessment (NEPSY-II), designed to assess the ability to judge line orientation. The Arrows subtest-level scores range from 1-19, with a low score indicating poor visuospatial skills, while a high score indicates excellent visuospatial skills.
Visual-spatial processing and mental rotation | Initial assessment and Follow-up assessment (6-8 weeks after Initial assessment)
  The Geometric Figures subtest of the revision of A Developmental Neuropsychological Assessment (NEPSY-II), designed to assess mental rotation, visuospatial analysis, and attention to detail. The Geometric Figures subtest-level scores range from 1-19, with a low score indicating difficulty with visuospatial perception, including mental rotation and with a high score indicating excellent visuospatial perception.
Selective visual attention | Initial assessment and Follow-up assessment (6-8 weeks after Initial assessment)
  The Cancellation subtest of the revision of the Wechsler Intelligence Scale for Children (WISC-IV), designed to measure processing speed. The Raw Score is converted to a Scaled Score (1-19), which is converted to a Percentile Rank. The higher the raw score, the higher the Scaled Score, and the Percentile Rank. The higher the score, the better the visual processing speed.
Visual-spatial decision making and visual-motor speed | Initial assessment and Follow-up assessment (6-8 weeks after Initial assessment)
  Coding subtest of the revision of the Wechsler Intelligence Scale for Children (WISC-IV), designed to measure visual-motor speed and complexity and motor coordination. The Raw Score is converted to a Scaled Score (1-19), which is converted to a Percentile Rank. The higher the raw score, the higher the Scaled Score, and the Percentile Rank. The higher the score, the better the visual-spatial and visual-motor skills.
Fine motor dexterity | Initial assessment and Follow-up assessment (6-8 weeks after Initial assessment)
  The Purdue Pegboard test, designed to measure manual dexterity and bimanual coordination.The test is comprised of 5 scores, each of the subtests are timed. Scores are continuous, the higher the score the greater the subjet's manual dexterity and bimanual coordination.
Visual-motor control | Initial assessment and Follow-up assessment (6-8 weeks after Initial assessment)
  The Visuomotor Precision subtest of the revision of A Developmental Neuropsychological Assessment (NEPSY-II), designed to assess graphomotor speed and accuracy. The Visuomotor Precision subtest-level scores range from 1-19, with a low score indicating difficulty with visuomotor control and with a high score indicating excellent visuomotor skills.
Neuroanatomical alterations in brain tissue structure | Baseline MRI and Follow-up MRI (6-8 weeks after Baseline MRI)
  Diffusion Tensor Imaging (DTI) scan: a spin-echo EPI DTI sequence (FOV = 240 x 240 mm, matrix = 96 x 96, in-plane resolution = 2.5 x 2.5 mm, slice thickness = 2.5 mm, number of slices =76, TR/TE = 9400/93.2 msec; sense factor = 2; NEX = 2). DTI measures anisotropic diffusion properties via diffusion indices.

SECONDARY OUTCOMES:
Adherence to the training plan | 6 weeks
  Adherence to the training plan will be evaluated using performance data collected by the apps. If performance data is not available from the apps, the participants will be given an activity log to record their usage time, games played, and scores obtained. Eighty-percent completion of the recommended time (24 hrs = 6 wks x 4 days/wk x 1 hr/day) is the goal of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Karen L Harpster, PhD, OTR/L, Principal Investigator — Children's Hospital Medical Center, Cincinnati